CLINICAL TRIAL: NCT07132892
Title: Clinical Use of Poly-4-Hydroxybutyrate Scaffold in Rhytidectomy- A Pilot Study
Brief Title: Poly-4-Hydroxybutyrate Scaffold in Rhytidectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey M. Kenkel (Other)
Responsible Party: Sponsor-Investigator, Jeffrey M. Kenkel, Chairman and Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU20251603
Record Dates: First submitted 2025-08-05; First posted 2025-08-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-08

CONDITIONS: Tissue Adhesion
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Intervention Model Description: Study procedure will be used to assess changes of the tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Healthy Participants (Experimental): Healthy subjects who received an elective rhytidectomy
  The GalaFLEX LITE is a surgical mesh scaffold composed of poly-4-hydroxybutyrate (P4HB) developed to prolong strength retention and reinforce soft tissue in patients undergoing plastic and reconstructive surgery.
  Interventions: Device: Galaflex Lite Scaffold

INTERVENTIONS:
Device: Galaflex Lite Scaffold — The GalaFLEX LITE is a surgical mesh scaffold composed of poly-4-hydroxybutyrate (P4HB) developed to prolong strength retention and reinforce soft tissue in patients undergoing plastic and reconstructive surgery.

SUMMARY:
The study is being conducted to objectively assess tissue changes following the use of P4HB in rhytidectomy to understand how the utilization of the surgical mesh may affect tissue mechanical strength and elasticity, wound healing, and scar formation dynamics.

DETAILED DESCRIPTION:
This is a prospective study designed to follow six (6) qualified and consenting adults, 18-80 years of age scheduled for an elective rhytidectomy with the Principal Investigator (PI). Subjects will be evaluated at baseline, month 1, month 6 and month 12. The effects of the study device will be analyzed at all follow up visits through clinical/3D photography, non-invasive skin assessments and subject/physician questionnaires. The PI will be collecting tissue samples during their surgical procedure, month 6 and month 12 visits. Histopathology will be completed on the collected sample to assess changes of the tissue after the subjects rhytidectomy.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria

1. Healthy adults 18-80 years of age
2. Planned/scheduled rhytidectomy at UT Southwestern with the study doctor
3. Willing to return for follow up visits and undergo study evaluations

Exclusion Criteria

1. Individuals diagnosed with known reaction to device material (tetracycline hydrochloride, kanamycin sulfate, etc)
2. Individuals who have significant scarring on the test area
3. Individuals with a disorder to negatively affect wound healing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasonography | Baseline, Month 3 and Month 6 and Month 12
  Ultrasonography will be used to evaluate the skin thickness and density for research purposes.
Bio-mechanical Tissue Characterization | Baseline, Month 3 and Month 6 and Month 12
  BTC will be used to measure skins laxity, viscoelasticity deformation, stiffness, energy absorption, elasticity, and deformation values for research purposes.
  Change from baseline will be calculated to assess change

SECONDARY OUTCOMES:
Histological Assessment | Baseline, Month 6 and Month 12
  Tissue will be obtained, for research purposes, to assess histological evaluation assessment.
  Change from baseline will be calculated to assess change
Instron Biomedical Testing | Baseline, Month 6 and Month 12
  The Instron device measures the mechanical properties of the tissue.
Face-Q: Satisfaction with Facial Appearance | Baseline, Month 6 and Month 12
  scale that measures a patient's overall satisfaction with how their face looks. It assesses things like symmetry, harmony, proportion, and vitality.
  A scale that measures a patient's overall satisfaction with how their face looks. It assesses things like symmetry, harmony, proportion, and vitality.
  A score from 0 to 100, where a higher score indicates a better outcome or greater satisfaction
Face-Q: Satisfaction with Outcome | Baseline, Month 6 and Month 12
  A series of positively worded questions to ask patients directly how they feel about the outcome.
  A score from 0 to 100, where a higher score indicates greater satisfaction with the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No